CLINICAL TRIAL: NCT01096303
Title: Effects of Marijuana Smoking on Pulmonary Function in Patients With COPD
Brief Title: Effects of Marijuana Used on Lung Function in Persons With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Rosa Estrada Y Martin, Associate Professor - I/M Pulmonary and Critical Care, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-09-0362
Record Dates: First submitted 2010-03-24; First posted 2010-03-31 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; pulmonary function; tobacco and marihuana smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Marijuana Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD tobacco and/or marihuana users: COPD patients with history of tobacco and/or marihuana smoking.

SUMMARY:
The main hypothesis is that persons that smoke or smoked tobacco and marihuana have worsen lung function as compared with persons that only smoke or smoked tobacco.

DETAILED DESCRIPTION:
We will follow persons with already diagnosed COPD (chronic bronchitis and/or emphysema). Obtain their smoking history: tobacco and marihuana and review their pulmonary function study results. Then we are planning to compare both groups.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients former or current tobacco smokers
* COPD patients former or current tobacco and marihuana smokers

Exclusion Criteria:

* History of COPD without pulmonary function testing
* Refusal to provide smoking or marihuana used history

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients recruited in pulmonary clinic.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-11; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Obstructive limitation in pulmonary function test | 1 year
  Comparison on the severity of obstruction among both groups

SECONDARY OUTCOMES:
Decreased diffusion capacity for carbon monoxide | 1 year
  Comparison on the severity of decreased DLco among groups.
Airtrapping | 1 year
  Comparison on the severity of air-trapping by pulmonary function testing among groups.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Estrada-Y-Martin, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Lyndon B Johnson General Hospital, Houston, Texas
  - The University of Texas- Health Science Center at Houston, Houston, Texas